CLINICAL TRIAL: NCT02741401
Title: COMplementary Hand-foot Massage to Improve Experience of illneSs Trial
Acronym: COMMIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Principal Investigator, M.J.M.T. Wolters, Dr. J.H.M.B. Stoot, Zuyderland Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: COMMIS
Record Dates: First submitted 2016-04-04; First posted 2016-04-18 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Gastrointestinal Cancer
Keywords: Complementary therapies; Massage; Gastrointestinal cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

ARMS (2):
- Therapy standard (Active Comparator): Patients receive usual postoperative care
  Interventions: Other: Usual post-operative care
- Therapy standard + hand-foot massage (Experimental): Patients receive usual postoperative care and hand-foot massage
  Interventions: Other: Usual post-operative care; Other: Hand-foot massage

INTERVENTIONS:
Other: Usual post-operative care — Usual post-operative care concerning patients who underwent surgery because of gastrointestinal malignancy
Other: Hand-foot massage — Hand-foot massage administered during 5 consecutive days postoperatively by trained volunteers, concerning patients who underwent surgery because of gastrointestinal malignancy
  Arms: Therapy standard + hand-foot massage

SUMMARY:
The COMplementary hand-foot Massage to Improve experience of ilneSs trial (COMMIS trial) is a prospective, randomized trial and executed at a Western referral Centre: Zuyderland Medical Centre located Sittard-Geleen, The Netherlands concerning patients who underwent surgery for gastrointestinal malignancy. During 5 consecutive days, the intervention group received postoperatively hand-foot massage administered by trained volunteers.

The aim of this study is to investigate the effect of complementary therapies concerning quality of life, pain, nausea, fatigue, sleeping problems, mood and stress in patients who underwent an operation as a result of gastrointestinal malignancy (stomach or colorectal).

DETAILED DESCRIPTION:
The COMplementary hand-foot Massage to Improve experience of ilneSs trial (COMMIS trial) is a prospective, randomized trial and executed at a Western referral Centre: Zuyderland Medical Centre located Sittard-Geleen, The Netherlands.

The aim of this study is to investigate the effect of complementary therapies concerning quality of life, pain, nausea, fatigue, sleeping problems, mood and stress in patients who underwent an operation as a result of gastrointestinal malignancy (stomach or colorectal). Patients had to be >18 years of age. Exclusion criteria were patients who were not able to undergo massage, not able to sign informed consent or speaking the native language, deaf patients and patients having a hand- or foot disorder.

Primary outcome measure is quality of life, including psychological state, level of functioning in daily life and pain. Secondary outcome measures are patient satisfaction about the received hospital care and the need for complementary medicine.

Recruitment takes place during the second preoperative appointment at the clinic, where eligible patients receive oral and written information about the study. One week after this conversation, patients are asked if they are interested to participate. If so, informed consent is obtained and remaining questions are answered.

Randomization takes place by the randomization program ALEA. It was not possible to blind investigator, patient, physician or nurse.

Patient groups consist of an intervention group (51 patients) and a control group (51 patients). The intervention group receives postoperatively during 5 consecutive days hand-foot massage from volunteers who are trained by a professional. It was not possible to receive massage in the weekends because of the absence of the volunteers. The technique comprised standard 'Swedish' massage, which means applying kneading and strokes to soft tissues and muscles. The intervention was performed by applying ethereal oils from Volatile, which consisted of 10% jojoba and 90% almond oil.

The control group receives the usual care.

Patients from both groups are asked to fill in questionnaires about health status/health related quality of life (EQ-5D-3L) and anxiety/depression (HADS-NL) at specific moments in time. Those include one week pre-operatively (baseline), post-operative day (POD) 1, POD3, POD5 and when they return at the policlinic after hospital's discharge. Before discharge, every patient is asked to fill in a questionnaire about patient satisfaction concerning the received hospital care as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent an operation as a result of gastrointestinal malignancy (stomach or colorectal).
* Patients >18 years of age.

Exclusion Criteria:

* Patients who were not able to undergo massage
* Patients who were not able to sign informed consent
* Patients who did not speak the native language
* Deaf patients
* Patients having a hand- or foot disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in quality of life as assessed by EuroQol-5D-L3 (EQ-5D-L3) questionnaire | From day of surgery until policlinical visit after hospital's discharge assessed up to 4 weeks
  To assess health-related quality of life, patients were asked to fill in the short generic EQ-5D-L3 questionnaire. Patients have to fill in those questionnaires at certain moments in time, from the day of surgery until the first visit at the policlinic after hospital's discharge. Patients are hospitalized about 1-2 weeks and their first policlinical visit after discharge is most often set at 1-2 weeks. That's why the time frame is estimated at 4 weeks.
  This questionnaire comprises health-related quality of life questions, e.g. state of mobility, self-care, daily activities, mood and pain.
Change from baseline in anxiety and depression as assessed by Hospital Anxiety and Depression Scale (HADS) questionnaire | From day of surgery until policlinical visit after hospital's discharge assessed up to 4 weeks
  Anxiety and depression is measured by using the Hospital Anxiety and Depression Scale (HADS). Patients have to fill in those questionnaires at certain moments in time, from the day of surgery until the first visit at the policlinic after hospital's discharge. Patients are hospitalized about 1-2 weeks and their first policlinical visit after discharge is most often set at 1-2 weeks. That's why the time frame is estimated at 4 weeks.

SECONDARY OUTCOMES:
Patient satisfaction about the received hospital care and hand-foot massage (if applicable) as assessed by questionnaire | From day of surgery until hospital's discharge assessed up to 2 weeks
  Patients are asked to fill in a questionnaire about the received hospital care and hand-foot massage (if applicable) at hospital's discharge. Patients have to fill in this questionnaires at hospital's discharge. Patients are hospitalized for 1-2 weeks, which means that the estimated time frime would be about 2 weeks (from day of surgery until date of discharge). That's why the time frame is estimated at 2 weeks.
Patients' opinion and need about hand-foot massage's utility as assessed by questionnaire | From day of surgery until policlinical visit after hospital's discharge assessed up to 2 weeks
  Patients are asked to fill in a questionnaire about their opinion about receiving hand-foot massage at hospital's discharge, even if they themselves were not randomized in the intervention group. Patients have to fill in this questionnaires at hospital's discharge. Patients are hospitalized for 1-2 weeks, which means that the estimated time frime would be about 2 weeks (from day of surgery until date of discharge). That's why the time frame is estimated at 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jan H. Stoot, Dr., Principal Investigator — Zuyderland MC